CLINICAL TRIAL: NCT01079806
Title: A Comparative Study of the Antiviral Efficacy and Safety of Entecavir (ETV) Versus Placebo in Pediatric Subjects With Chronic Hepatitis B Virus (HBV) Infection Who Are HBeAg-Positive
Brief Title: A Phase III Study of the Safety and Efficacy of Entecavir in Pediatric Patients With Chronic Hepatitis B Virus Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI463-189 ST
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2019-04

CONDITIONS: Chronic Hepatitis B Virus, Pediatric
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Entecavir (Active Comparator): Participants received entecavir, 0.015 mg/kg up to 0.5 mg, once daily, for 96 to 144 weeks, depending on response
  Interventions: Drug: Entecavir
- Placebo (Placebo Comparator): Participants received placebo, 0 mg, once daily, for 48 to 96 weeks, depending on response
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Entecavir — Tablets/oral solution, 0.015 mg/kg up to 0.5 mg, administered orally, once daily, for 96 to144 weeks, depending on response
  Other Names: Baraclude; BMS-200475
  Arms: Entecavir
Drug: Placebo — Tablets/oral solution, 0 mg, administered orally, once daily, for 48 to 96 weeks, depending on response
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of entecavir in pediatric patients with chronic hepatitis B virus infection

ELIGIBILITY:
Key Inclusion Criteria

* Males and females, aged 2 to <18 years
* Hepatitis B surface antigen-positive
* Detectable hepatitis B e (HBe) antigen, and no detectable anti-HBe antibodies
* Alanine aminotransferase (ALT) 1.5 to <10 times the upper limit of normal at screening and within 8 to 24 weeks prior to screening
* Evidence of the presence of hepatitis B virus DNA at least 4 weeks before screening and >100,000 copies/mL at screening

Key Exclusion Criteria

* Any prior therapy with entecavir
* At least 12 weeks of prior therapy with any nucleoside or nucleotide antiviral agent
* Therapy with interferon alpha, thymosin alpha, or nucleototide antiviral agents within 24 weeks of screening
* Coinfection with HIV, hepatitis C virus, or hepatitis D virus
* Decompensated liver disease
* Liver transplant recipients
* Other forms of acute and chronic conditions which may cause increased ALT levels
* Children who were breastfed while their mothers received lamivudine or whose mothers received lamivudine during pregnancy

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2010-06-30 (Actual); Primary Completion 2013-03-31 (Actual); Study Completion 2018-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (42):
- United States (15):
  - University Of California, San Francisco, San Francisco, California
  - Connecticut Children'S Medical Center, Hartford, Connecticut
  - Children'S National Medical Center, Washington D.C., District of Columbia
  - University Of Florida, Gainesville, Florida
  - Romero, Rene, Atlanta, Georgia
  - Indiana University School Of Medicine / Riley Hospital, Indianapolis, Indiana
  - Johns Hopkins School Of Medicine, Baltimore, Maryland
  - Shah, Uzma, Boston, Massachusetts
  - Boston Childrens Hospital, Boston, Massachusetts
  - Mount Sinai Medical Center, New York, New York
  - Levine Children'S Hospital At Carolinas Medical Center, Charlotte, North Carolina
  - Children'S Hospital Of Philadelphia, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Texas Children'S Hospital, Houston, Texas
  - Inova Fairfax Hospital For Children, Fairfax, Virginia
- Local Institution, Bunos Aires, Buenos Aires, Argentina
- Local Institution, Brussels, Belgium
- Local Institution, Toronto, Ontario, Canada
- Germany (3):
  - Local Institution, Mainz, Rhineland-Palatinate
  - Local Institution, Starnberg
  - Local Institution, Wuppertal
- Local Institution, Thesaloniki, Greece
- India (2):
  - Local Institution, Guwahati
  - Local Institution, Hyderabad
- Israel (3):
  - Local Institution, Beersheba
  - Local Institution, Petah Tikva
  - Local Institution, Safed
- Poland (3):
  - Local Institution, Bydgoszcz
  - Local Institution, Krakow
  - Local Institution, Wroclaw
- Romania (3):
  - Local Institution, Bucharest
  - Local Institution, Iași
  - Local Institution, Timișoara
- Russia (3):
  - Local Institution, Moscow
  - Local Institution, Novokuznetsk
  - Local Institution, Saint Petersburg
- South Korea (2):
  - Local Institution, Daegu
  - Local Institution, Seoul
- Taiwan (2):
  - Local Institution, Tainan
  - Local Institution, Taipei
- United Kingdom (2):
  - Local Institution, London, Greater London
  - Local Institution, Birmingham, West Midlands

REFERENCES:
- [Derived] Jonas MM, Chang MH, Sokal E, Schwarz KB, Kelly D, Kim KM, Ling SC, Rosenthal P, Oraseanu D, Reynolds L, Thiry A, Ackerman P. Randomized, controlled trial of entecavir versus placebo in children with hepatitis B envelope antigen-positive chronic hepatitis B. Hepatology. 2016 Feb;63(2):377-87. doi: 10.1002/hep.28015. Epub 2015 Oct 16. PMID 26223345
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 228 patients enrolled, 43 no longer met study criteria, 4 withdrew consent, and 1 withdrew for surgery. While the primary endpoint analysis was based on a randomized sample size of 123 participants, the overall study population was augmented to 180 to meet global regulatory requirements. All 180 randomized patients received study drug.
Period: Day 1 to Week 96
Arm/Group | Entecavir | Placebo
Started | 120 | 60
Received Treatment | 120 | 60
Primary Endpoint Cohort | 82 | 41
Completed | 113 | 53
Not Completed | 7 | 7
Not completed — Adverse Event | 0 | 3
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Pregnancy | 0 | 1
Not completed — Poor compliance or noncompliance | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Subject request to stop study treatment | 1 | 0
Not completed — Removal by Medical Monitor | 0 | 1
Period: Long-term Follow-up: Day 1-End of Study
Arm/Group | Entecavir | Placebo
Started (Entered from start to end of long-term follow-up) | 111 | 58
Completed | 92 | 43
Not Completed | 19 | 15
Not completed — Withdrawal by Subject | 13 | 8
Not completed — Investigator Left Institution | 0 | 1
Not completed — Lost to Follow-up | 6 | 6

BASELINE CHARACTERISTICS:
Population: All participants who received study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Entecavir | Placebo | Total
Number analyzed (Participants) | 120 | 60 | 180
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.5 (4.87) | 10.8 (4.82) | 10.6 (4.84)
Age, Customized [Number; unit: participants]
  >=2 years to <=6 years | 27 | 14 | 41
  >6 years to <=12 years | 31 | 15 | 46
  >12 years to <18 years | 62 | 31 | 93
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 29 | 71
  Male | 78 | 31 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 48 | 21 | 69
  Unknown or Not Reported | 70 | 39 | 109
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 57 | 30 | 87
  Black/African American | 14 | 2 | 16
  Native Hawaiian/Other Pacific Islander | 1 | 0 | 1
  White | 44 | 27 | 71
  Other | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a Combination of Hepatitis B Virus (HBV) DNA Suppression and Hepatitis B e Antigen (HBeAg) Seroconversion at Week 48
Description: Suppression=HBV DNA<50 IU/mL (approximately 300 copies/mL) using the Roche COBAS TaqMan HBV Test for use with the High Pure System assay; seroconversion=undetectable HBeAg and detectable anti-hepatitis B e antibodies. While the analysis of the primary endpoint was based on a randomized sample size of 123 participants (the Primary Cohort), the size of the overall study population was augmented to 180 randomized participants to meet global regulatory requirements.
Time Frame: At Week 48
Population: The first 123 participants who were randomized and received treatment (referred to as the Primary Cohort)
Measure: Number; unit: Percentage of participants
Arm/Group | Entecavir | Placebo
Number analyzed (Participants) | 82 | 41
Percentage of participants | 24.4 | 2.4
Statistical Analysis 1: Comparison: Entecavir vs Placebo; Test type: Superiority; p = 0.0049, Normal approximation; Difference estimate = 20.2, 95% CI 2-sided [9.1 to 31.4] — Difference estimate is stratified by age randomization strata, using Cochran-Mantel-Haenszel weighting

2. Secondary Outcome: Percentage of Participants With Hepatitis B Virus (HBV) DNA <50 IU/mL at Week 48
Description: While the analysis of the primary endpoint was based on a randomized sample size of 123 participants (the Primary Cohort), the size of the overall study population was augmented to 180 randomized participants to meet global regulatory requirements.
Time Frame: At Week 48
Population: The first 123 participants who were randomized and received treatment (referred to as the Primary Cohort)
Measure: Number; unit: Percentage of participants
Arm/Group | Entecavir | Placebo
Number analyzed (Participants) | 82 | 41
Percentage of participants | 46.3 | 2.4
Statistical Analysis 1: Comparison: Entecavir vs Placebo; Test type: Superiority; p < 0.0001, Normal approximation; Difference estimate = 41.8, 95% CI 2-sided [29.4 to 54.2] — Difference estimate is stratified by age randomization strata, using Cochran-Mantel-Haenszel weighting

3. Secondary Outcome: Percentage of Participants With Serum Alanine Aminotransferase ≤1*Upper Limit of Normal at Week 48
Description: as for outcome 2
Time Frame: At Week 48
Population: The first 123 participants who were randomized and received treatment (referred to as the Primary Cohort)
Measure: Number; unit: Percentage of participants
Arm/Group | Entecavir | Placebo
Number analyzed (Participants) | 82 | 41
Percentage of participants | 67.1 | 22.0
Statistical Analysis 1: Comparison: Entecavir vs Placebo; Test type: Superiority; p < 0.0001, Normal approximation; Difference estimate = 45.2, 95% CI [29.2 to 61.2] — Difference estimate is stratified by age randomization strata, using Cochran-Mantel-Haenszel weighting

4. Secondary Outcome: Percentage of Participants With Hepatitis B Virus DNA <Limit of Quantitation (LOQ) at Week 48
Description: LOQ=29 IU/mL. While the analysis of the primary endpoint was based on a randomized sample size of 123 participants (the Primary Cohort), the size of the overall study population was augmented to 180 randomized participants to meet global regulatory requirements.
Time Frame: At Week 48
Population: The first 123 participants who were randomized and received treatment (referred to as the Primary Cohort)
Measure: Number; unit: Percentage of participants
Arm/Group | Entecavir | Placebo
Number analyzed (Participants) | 82 | 41
Percentage of participants | 42.7 | 2.4
Statistical Analysis 1: Comparison: Entecavir vs Placebo; Test type: Superiority; p < 0.0001, Normal approximation; Difference estimate = 38.2, 95% CI 2-sided [25.9 to 50.5] — Difference estimate is stratified by age randomization strata, using Cochran-Mantel-Haenszel weighting

5. Secondary Outcome: Percentage of Participants With Hepatitis B e Antigen (HBeAg) Seroconversion at Week 48 (Undetectable HBeAg and Presence of Anti-HBeAb)
Description: Percentage of participants in the primary cohort with HBeAg seroconversion (undetectable HBeAg and presence of anti-HBe antibodies) at week 48
Time Frame: At Week 48
Population: The first 123 participants who were randomized and received treatment (referred to as the Primary Cohort)
Measure: Number; unit: Percentage of participants
Arm/Group | Entecavir | Placebo
Number analyzed (Participants) | 82 | 41
Percentage of participants | 24.4 | 12.2
Statistical Analysis 1: Comparison: Entecavir vs Placebo; Test type: Superiority; p = 0.11, Normal approximation; Difference estimate = 12.1, 95% CI 2-sided [-1.5 to 25.7] — Difference estimate is stratified by age randomization strata, using Cochran-Mantel-Haenszel weighting

6. Secondary Outcome: Percentage of Participants Who Achieved Sustained HBeAg Seroconversion During Off-treatment Follow up Among Participants Who Achieved HBeAg Seroconversion at End of Dosing (EOD).
Description: Participants who demonstrated HBeAg seroconversion at EOD were followed and assessed for presence of sustained HBeAg seroconversion during entire study. The study reached the end of dosing (EOD) on 22 Feb-2016.
Time Frame: Week 48, EOD (2 years)
Population: Participants who achieved HBeAg seroconversion at end of treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Entecavir | Placebo
Number analyzed (Participants) | 39 | 22
Percentage of participants
  EOD (end of dosing) | 100.0 | 100.0
  Week 48 | 74.4 | 59.1

7. Secondary Outcome: Number of Participants With Adverse Events (Including Palatability Issues), SAEs, Discontinuous Due to Adverse Events, and HBV Disease Progression Through Week 48
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Related=having certain, probable, possible, or unknown relationship to study drug. Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening or disabling, Grade 5=Death. ALT=alanine aminotransferase.
Time Frame: Day 1 through Week 48 on blinded therapy
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Entecavir | Placebo
Number analyzed (Participants) | 120 | 60
participants
  Deaths | 0 | 0
  Serious Adverse Events | 4 | 7
  Discontinuation due to Adverse Event | 0 | 2
  any adverse event | 78 | 46
  Related Adverse Events | 11 | 6
  Related Grade 2 - 4 Adverse Events | 4 | 2
  Grade 3 - 4 Adverse Events | 4 | 3
  ALT Flares | 2 | 5
  HBV disease progression | 0 | 0
  Malignant neoplasms or pre-malignant lesions | 0 | 0

8. Secondary Outcome: Number of Participants With Laboratory Test Results Meeting the Criteria for Abnormality (Grades 1-4)
Description: Toxicities graded per Division of AIDS criteria, Version 1.0, and modified World Health Organization criteria. INR=international normalization ratio of prothrombin time; ULN=upper limit of normal. Hemoglobin (g/dL): Grade 1=10-10.9; Grade 2=9-9.9; Grade 3=7-8.9; Grade 4= <7. Platelets (/mm^3): Grade 1=100,000-124,999; Grade 2=50,000-99,999; Grade 3=25,000-49,999; Grade 4= <25,000. INR (*ULN): Grade 1=1.1-1.5; Grade 2=1.6-2; Grade 3=2.1-3; Grade 4= >3. WBC (/mm^3): Grade 1=2000-2500; Grade 2=1500-1999; Grade 3=1000-1499; Grade 4= <1000. Neutrophils (/mm^3): Grade 1=1000-1300; Grade 2=750-999; Grade 3=500-749; Grade 4= <500.
Time Frame: Day 1 through Week 48 on blinded therapy
Population: All treated subjects
Measure: Number; unit: Participants
Arm/Group | Entecavir | Placebo
Number analyzed (Participants) | 120 | 60
Participants
  Hemoglobin: number analyzed (Participants) | 119 | 60
  Hemoglobin | 5 | 4
  Platelets: number analyzed (Participants) | 119 | 60
  Platelets | 3 | 2
  INR: number analyzed (Participants) | 117 | 59
  INR | 2 | 6
  White blood cells (WBC): number analyzed (Participants) | 119 | 60
  White blood cells (WBC) | 2 | 1
  Neutrophils + bands (absolute): number analyzed (Participants) | 119 | 60
  Neutrophils + bands (absolute) | 14 | 2

9. Secondary Outcome: Number of Participants With Laboratory Test Results Meeting the Criteria for Abnormality (Grades 1-4) (Continued)
Description: Toxicities graded per Division of AIDS criteria, Version 1.0, and modified World Health Organization criteria. ALT=alanine aminotransferase; AST=aspartate aminotransferase; BUN=blood urea nitrogen; ULN=upper limit of normal; LLN=lower limit of normal. ALT, AST (*ULN): Grade 1=1.25-2; Grade 2=2.6-5; Grade 3=5.1-10; Grade 4 => 10. Bilirubin (*ULN): Grade 1 = 1.1-1.5; Grade 2=1.6-2.5; Grade 3 = 2.6-5; Grade 4= >5. Albumin (g/dL): Grade 1=3- <LLN; Grade 2=2-2.9; Grade 3= <2. Lipase (*ULN): Grade 1=1.1-1.5; Grade 2=1.6-3; Grade 3=3.1-5; Grade 4= >5. BUN/urea (*ULN): Grade 1=1.25-<2.6; Grade 2=2.6-<5.1; Grade 3=5.1-10; Grade 4= >10. Chloride, high (mEq/L): Grade 1=113-<117; Grade 2=117-<121; Grade 3=121-125; Grade 4= >125. Potassium, low (mEq/L): Grade 1=3-3.4; Grade 2=2.5-<3; Grade 3=2-<2.5; Grade 4=<2. Potassium, high (mEq/L): : Grade 1= 5.6-<6.1; Grade 2=6.1-<6.6; Grade 3=6.6-7; Grade 4= >7. Sodium, high (mEq/L): Grade 1=146<151; Grade 2=151-<155; Grade 3=155-<160; Grade 4= >=160.
Time Frame: Day 1 through Week 48 on blinded therapy
Population: All randomized participants who received at least 1 dose of study medication
Measure: Number; unit: participants
Arm/Group | Entecavir | Placebo
Number analyzed (Participants) | 120 | 60
participants
  ALT: number analyzed (Participants) | 119 | 60
  ALT | 113 | 59
  AST: number analyzed (Participants) | 119 | 60
  AST | 87 | 51
  Total bilirubin: number analyzed (Participants) | 119 | 60
  Total bilirubin | 5 | 6
  Albumin: number analyzed (Participants) | 119 | 60
  Albumin | 0 | 1
  Lipase: number analyzed (Participants) | 119 | 60
  Lipase | 38 | 20
  BUN/Urea: number analyzed (Participants) | 119 | 60
  BUN/Urea | 10 | 2
  Chloride, high: number analyzed (Participants) | 119 | 60
  Chloride, high | 2 | 1
  Potassium, low: number analyzed (Participants) | 119 | 60
  Potassium, low | 1 | 1
  Potassium, high: number analyzed (Participants) | 119 | 60
  Potassium, high | 1 | 0
  Sodium, high: number analyzed (Participants) | 119 | 60
  Sodium, high | 8 | 4

10. Secondary Outcome: Percentage of Participants With HBeAg Seroconversion on ETV Over-time at Week 96 (All ETV Cohort)
Description: HBe seroconversion=undetectable HBe antigen and detectable anti-HBe antibodies. While the analysis of the primary endpoint was based on a randomized sample size of 123 participants (the Primary Cohort), the size of the overall study population was augmented to 180 randomized participants to meet global regulatory requirements.
Time Frame: At Week 96
Population: Randomized ETV subjects combined with PBO-randomized participants who received open-label ETV
Measure: Number; unit: Percentage of participants
Groups:
- Blinded and Open-Label (All ETV): Randomized ETV subjects combined with PBO-randomized subjects who received open-label ETV
Arm/Group | Blinded and Open-Label (All ETV)
Number analyzed (Participants) | 171
Percentage of participants | 38.6

11. Secondary Outcome: Percentage of Participants Who Maintained HBeAg Seroconversion at Week 96 (End of Blinded Therapy) Among Participants With HBeAg Seroconversion at Week 48
Description: Participants who achieved HBeAg seroconversion by Week 48 and maintained seroconversion to week 96
Time Frame: At Week 96
Population: participants with HBeAg seroconversion at Week 48
Measure: Number; unit: Percentage of participants
Arm/Group | Entecavir | Placebo
Number analyzed (Participants) | 120 | 60
Percentage of participants
  Week 48 | 24.2 | 10.0
  Week 96: number analyzed (Participants) | 120 | 50
  Week 96 | 36.7 | 20.0

12. Secondary Outcome: Percentage of Participants With Death as Outcome, Serious Adverse Events (SAEs), Discontinuations Due to Adverse Events (AEs), Related AEs, Grade 2-4 Related AEs, Grade 3-4 AEs, Malignancies, ALT Flares, and Hepatic Disease Progression Through Week 96
Description: as for outcome 7
Time Frame: Day 1 through Week 96
Population: All treated participants
Measure: Number; unit: Percentage of participants
Groups:
- Blinded and Open-Label (All ETV): All ETV group during long-term follow-up that show increased ALT (alanine aminotransferase)
Arm/Group | Blinded and Open-Label (All ETV)
Number analyzed (Participants) | 171
Percentage of participants
  Deaths | 0
  SAEs | 4.7
  Discontinuations due to AEs | 0.6
  Related AEs | 8.2
  Grade 2-4 Related AEs | 2.3
  Grade 3-4 AEs | 4.1
  Malignancies | 0
  ALT flares | 1.8
  Hepatic disease progression | 0

13. Secondary Outcome: Percentage of Participants With HBeAg Seroconversion (Undetectable HBeAg and Presence of Anti-HBeAb) up to Week 96
Description: On Treatment through week 96 - 2 year cohort NC = F: (The numerator was based on participants meeting the response criteria. The denominator was based on treated participants. Participants who had missing data at the analysis week were considered failures.)
Time Frame: up to week 96
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Entecavir
Number analyzed (Participants) | 120
Percentage of participants | 40.8

14. Secondary Outcome: Histological Analysis (Percentage) Among Participants With Available Liver Biopsy Data
Description: Liver function test elevations and abnormalities on blinded and open-label ETV (the All ETV Safety Cohort). Participants who experienced elevation of alanine aminotransferase (ALT) greater than three times ETV (entecavir) baseline measure (Participants who displayed liver biopsy with ALT value greater than three times baseline.)
Time Frame: Between weeks 48 and 96
Population: Randomized ETV subjects combined with PBO-randomized participants who received open-label ETV
Measure: Number; unit: Percentage of participants
Arm/Group | Blinded and Open-Label (All ETV)
Number analyzed (Participants) | 171
Percentage of participants | 5.9

15. Secondary Outcome: Percentage of Participants With HbeAg Loss at Weeks 48 and 96
Description: HBeAg Loss (NC = F and NC = M) - On Treatment through Week 96 - Year 2 Efficacy Cohort Non-Completer - Failure (NC=F): The numerator was based on participants meeting the response criteria. The denominator was based on treated participants. Participants who had missing data at the analysis week were considered failures. Non-Completer - Missing (NC=M): The numerator was based on participants meeting the response criteria. The denominator was based on participants with data at the analysis week. Participants who had missing data at the analysis week were excluded.
Time Frame: At 48 and 96 weeks
Population: Participants with response rates at weeks 48 and 96 in Entecavir (ETV) and Placebo (PBO) randomized cohort
Measure: Number; unit: Percentage of participants
Arm/Group | Entecavir | Placebo
Number analyzed (Participants) | 120 | 60
Percentage of participants
  48 weeks | 25.0 | 10.0
  96 Weeks: number analyzed (Participants) | 120 | 0
  96 Weeks | 40.8 |

ADVERSE EVENTS:
Time Frame: All non-serious adverse events were collected from start of study treatment through Week 48, while all serious adverse events were evaluated through out the study (5 years).
Groups:
- ETV (Entecavir): Subjects received 0.015 milligram per kilogram per day (mg/kg/day) (up to a maximum dose of 0.5 mg/day) ETV as oral solution or tablets, once daily (QD).
- PLACEBO: Subjects received ETV matched placebo as oral solution or tablets, QD.
Arm/Group | ETV (Entecavir) | PLACEBO
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/60
Serious Adverse Events (participants affected / at risk) | 4/120 | 9/60
Other Adverse Events (participants affected / at risk) | 76/120 | 45/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ETV (Entecavir) (N=120) | PLACEBO (N=60)
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 2
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Chronic hepatitis b (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 1 | 0
Infectious colitis (Infections and infestations) | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ETV (Entecavir) (N=120) | PLACEBO (N=60)
Abdominal discomfort (Gastrointestinal disorders) | 5 | 3
Abdominal pain (Gastrointestinal disorders) | 9 | 9
Diarrhoea (Gastrointestinal disorders) | 7 | 7
Dyspepsia (Gastrointestinal disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 6 | 5
Vomiting (Gastrointestinal disorders) | 14 | 10
Fatigue (General disorders) | 3 | 5
Pyrexia (General disorders) | 18 | 10
Bronchitis (Infections and infestations) | 8 | 6
Ear infection (Infections and infestations) | 7 | 1
Gastroenteritis (Infections and infestations) | 6 | 4
Influenza (Infections and infestations) | 6 | 4
Nasopharyngitis (Infections and infestations) | 18 | 14
Pharyngitis (Infections and infestations) | 5 | 11
Pharyngitis streptococcal (Infections and infestations) | 4 | 4
Pneumonia (Infections and infestations) | 6 | 0
Tonsillitis (Infections and infestations) | 6 | 1
Upper respiratory tract infection (Infections and infestations) | 19 | 12
Headache (Nervous system disorders) | 18 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Acne (Skin and subcutaneous tissue disorders) | 3 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 5
Rash (Skin and subcutaneous tissue disorders) | 7 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-12-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT01079806/SAP_000.pdf
  • Study Protocol (2012-09-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT01079806/Prot_001.pdf